CLINICAL TRIAL: NCT04541550
Title: An Open-label, Dose-escalation Study to Evaluate the Use of Allogeneic Micronized Amniotic Membrane Product for the Treatment of Hidradenitis Suppurativa
Brief Title: Allogeneic Micronized Amniotic Membrane Product for the Treatment of Hidradenitis Suppurativa
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study didn't proceed to FDA submission
Sponsor: IntegoGen, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT-001
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose AMP-001 (Experimental): 12.5 mg AMP-001 in 3 ml Saline
  Interventions: Drug: AMP-001 Low Dose
- Medium Dose AMP-001 (Experimental): 25 mg AMP-001in 3 ml Saline
  Interventions: Drug: AMP-001 Medium Dose
- High Dose AMP-001 (Experimental): 50 mg AMP-001 in 3 ml Saline
  Interventions: Drug: AMP-001 High Dose

INTERVENTIONS:
Drug: AMP-001 Low Dose — AMP-001, is manufactured from the amniotic membrane of the placenta and does not contain living cells.
  Other Names: 12.5 mg AMP-001
  Arms: Low Dose AMP-001
Drug: AMP-001 Medium Dose — AMP-001, is manufactured from the amniotic membrane of the placenta and does not contain living cells.
  Other Names: 25 mg AMP-001
  Arms: Medium Dose AMP-001
Drug: AMP-001 High Dose — AMP-001, is manufactured from the amniotic membrane of the placenta and does not contain living cells.
  Other Names: 50 mg AMP-001
  Arms: High Dose AMP-001

SUMMARY:
This study is an open-label, dose-escalation study enrolling 15 participants.

There are 3 cohorts:

1. Cohort I: 5 subjects each receiving 1 injection of IGN-AMP001 (12.5mg AMP-001 in 3ml Saline)
2. Cohort II: 5 subjects each receiving 1 injection of IGN-AMP001 (25 mg AMP-001 in 3 ml Saline)
3. Cohort III: 5 subjects each receiving 1 injection of IGN-AMP001 (50 mg AMP-001 in 3 ml Saline).

DETAILED DESCRIPTION:
Hidradenitis Suppurativa (HS) is a chronic inflammatory skin disease characterized by recurrent deep-seated boil-like abscesses and tracts under the skin. The most severe HS lesions are characterized by chronic non-healing sinuses, which form a wound-like environment as the abscesses heal; they produce significant skin scarring. Transcriptomic analysis of lesioned skin from HS patients suggests that it has similar pathology to other chronic wounds. IntegoGen's investigational product, IGN-AMP001, is manufactured from the amniotic membrane of the human placenta. The amnion membrane contains various cytokines and growth factors that promote wound healing. Local application of micronized dehydrated amnion membrane has been shown effective in treating chronic refractory non-healing dermal wounds of various etiologies in randomized clinical trials and case studies, which suggests it might be effective in treating HS wounds as well. Patients treated with IGN-AMP001 within IntegoGen associated clinics and other regenerative clinics have indicated positive responses. This study is designed to evaluate the safety, tolerability, and potential efficacy of IGN-AMP001 for HS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Can understand the nature of the procedure, and provide, or have a legal representative provide, a written informed consent.
* Clinically diagnosed with Hidradenitis Suppurativa characterized as Hurley Score, Stage II or Stage III.
* History of standard-of-care supportive treatment failure with corticosteroids and/or antibiotics within 30 days before the baseline visit.
* Must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at the baseline visit.
* No prior history of a biologic product or Humira for the treatment of Hidradenitis Suppurativa.

Exclusion Criteria:

* Intolerance or unwillingness to participate in all procedure(s) or medication(s) required of this protocol.
* Diagnosis or reported history of any of the folding conditions:

  1. Uncontrolled Diabetes Mellitus (HbA1c ≥9);
  2. Severe Morbid Obesity (BMI≥40);
  3. Chronic heart, renal, or hepatic disease;
  4. Neurodegenerative debilitating conditions, and
  5. Cancer.
* The participant is currently receiving or has received within 3 months before enrollment, medications or treatments that are known to affect the wound healing process, including but not limited to: chronic systemic steroid intake, history of recent changes in the participant's tissue integrity (i.e., thin, fragile skin with multiple hematomas or previous lacerations), current use of immune-suppressive drugs, radiation therapy, immunomodulating medications, and chemotherapy.
* The participant has received HS micronized amnion therapy in the last 90 days.
* Systolic blood pressure greater than 190 or less than 90 mmHg.
* Diastolic blood pressure greater than 105 or less than 50 mmHg.
* Early, symptomatic autonomic dysfunction.
* Abuse of prescription drugs, illegal substances, and/or alcohol.
* Females who are pregnant, nursing, or of childbearing potential and not using a reliable birth control method (such as, female use of a diaphragm, intrauterine device (IUD), or contraceptive sponge or gels, in addition to male use of a condom) or the female should be using prescribed "birth control" pills, injections, or implants. or who intend to become pregnant during their participation in the study.
* Clinically significant abnormal laboratory values at the time of the screening or baseline visit.
* Exposure to the investigational product within 3 months prior to enrollment or anticipate participation in any other investigational drug study or other interventional studies while enrolled in the study.
* In the opinion of the Principal Investigator, the participant should not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Total number of Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Mahoney, MD, Principal Investigator — West Houston Dermatology Laser and Skin Care Center
Locations (1):
- West Houston Dermatology Laser and Skin Care Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No